CLINICAL TRIAL: NCT01492192
Title: Prospective Study of 18F-RGD PET-CT in Assessment of Response to Antiangiogenic Treatment in Patients With Cancer and Comparison With Perfusion CT
Brief Title: RGD-PET-CT in Cancer Angiogenesis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: GE Healthcare (Industry); University of Oxford (Other)
Responsible Party: Principal Investigator, Linda Ward, Quality Manager, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EP-TSC-663; 2011-002833-20 (EudraCT Number)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Carcinoma, Renal Cell
Keywords: Angiogenesis; PET-CT; Perfusion-CT
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — AH 111585

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RCC Patients Antiangiogenic treatment (Experimental)
  Interventions: Drug: 18F-RGD-PET-CT and perfusion CT scans on 3 occasions

INTERVENTIONS:
Drug: 18F-RGD-PET-CT and perfusion CT scans on 3 occasions — Fluciclatide (GE Healthcare) (AH111585) is a small cyclic peptide containing the RGD tripeptide (figure 1), which preferentially binds with high affinity to α¬vβ3 integrins that are up-regulated in angiogenesis.
  The IMP is supplied as a solution for injection, 400 MBq at the reference date and time. Participants will receive one injection of the imaging agent at this dose on 3 occasions
  Other Names: αvβ3 Integrin Imaging with Fluciclatide (AH111585)

SUMMARY:
The goal of this clinical research study is to look at 2 new methods of scanning and see whether they can help researchers predict which tumours will respond to drugs that attack tumour blood supply.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should have advanced or metastatic RCC confirmed by histological diagnosis
2. Patients considered suitable for therapy with TKI for RCC according to responsible clinician
3. Measurable tumour according to RECIST v1.1 criteria
4. Standard staging CT scan performed within 28 days of first research scan
5. The patient has not received chemotherapy, radiotherapy, surgery or any other treatment against cancer within 4 weeks prior to recruitment
6. Age ≥18 years
7. Adequate renal function (creatinine <1.25xULN)
8. Patient is able to tolerate and comply with scanning procedure
9. Patient is not lactating or pregnant
10. Absence of any psychological, familial, sociological or geographical condition which in the opinion of the Investigator may potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
11. Able and willing to give informed consent

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in tumour uptake of the fluciclatide imaging agent | Prior to starting anti-angiogenic treatment, repeat after ~4 and 16 weeks of treatment
  % change in SUVmax

SECONDARY OUTCOMES:
Tumour response within an individual patient | Prior to starting anti-angiogenic treatment, repeat after ~4 and 16 weeks of treatment
  % change in size
Changes of kinetic parameters on CT perfusion imaging | Prior to starting anti-angiogenic treatment, repeat after ~4 and 16 weeks of treatment
  BV, BF and Ki
Absolute and relative tumour uptake and retention of fluciclatide | Prior to starting anti-angiogenic treatment, repeat after ~4 and 16 weeks of treatment
Progression free survival at 12 months- | 12 months after the final reseach scan.
  Time from last study scan to the date of disease progression or death due to the disease,whichever occurs first.
Overall survival at 12 months | 12 months after the final reseach scan.
Safety profile | within 12 months of the last research scan
  Number of participants with adverse events attributed to the 18F-RDG-PET imaging agent (CTCAE Criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Gleeson, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Department of Radiology, Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom